CLINICAL TRIAL: NCT07208214
Title: A Randomised Parallel-group Study of Texture and Colour Enhancement Imaging (TXI) Versus Dye Chromoendoscopy for Dysplasia Detection in IBD Surveillance.
Brief Title: Texture and Colour Enhancement Imaging (TXI) Versus Dye Chromoendoscopy for Dysplasia Detection in IBD Surveillance.
Acronym: TXIorDyE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD24/053
Record Dates: First submitted 2025-09-17; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: IBD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TXI (Active Comparator): Participants allocated to the "TXI" group undergo withdrawal using Texture and Colour Enhancement Imaging
  Interventions: Diagnostic Test: TXI
- Dye (Other): Participants allocated in the "Dye" group receive withdrawal with Dye chromoendoscopy.
  Interventions: Diagnostic Test: TXI

INTERVENTIONS:
Diagnostic Test: TXI — Participants allocated to the "TXI" group undergo withdrawal using Texture and Colour Enhancement Imaging, while those in the "Dye" group receive withdrawal with Dye chromoendoscopy. Both procedures follow standardized protocols outlined in the study design.

SUMMARY:
In individuals with inflammatory bowel disease (IBD), bowel cancer can develop from abnormal cell changes (dysplasia). Regular colonoscopies are recommended to identify these early changes, which can be difficult to detect because they are often small and subtle. Dye-based imaging has been used to improve detection, but it requires additional preparation and time. Texture and Colour Enhancement Imaging (TXI) is a newer method available in clinical practice that adjusts brightness, colour, and texture on high-definition cameras. This study will compare TXI with dye-based imaging to assess which approach detects precancerous changes more effectively in patients with IBD.

DETAILED DESCRIPTION:
Bowel cancer in individuals with inflammatory bowel disease (IBD) often develops from abnormal changes in the cells lining the bowel, known as dysplasia. International guidelines recommend undertaking regular colonoscopies to check for precancerous changes in patients with IBD. In the past, these precancerous changes were thought to be invisible, but with improved camera imaging technology, most cases of early changes can now be detected. However, early precancerous changes remain difficult to identify because they often appear as small, flat, and subtle lesions.

Studies have shown that applying dye to the bowel lining during colonoscopy can improve the detection of early changes compared with standard endoscopy. Nevertheless, the use of dye presents challenges, including additional preparation, longer procedure time, and the need for specific training. Newer high-definition cameras have demonstrated higher detection rates than older standard cameras. Advances in imaging technology have also led to the development of novel techniques designed to improve detection and identification of abnormal tissues. One such technique is Texture and Colour Enhancement Imaging (TXI), which enhances texture, brightness, and colour in high-definition cameras, making small and subtle differences in tissue more visible. This technology is now available in routine clinical practice with the EVIS X1 system (Olympus).

No randomized studies have yet evaluated the effectiveness of TXI in detecting early precancerous changes during colonoscopy in patients with IBD. The present study is designed to compare TXI with dye-based imaging in order to determine which method more effectively detects precancerous changes in IBD.

ELIGIBILITY:
Inclusion Criteria:

* Patients >16 with inflammatory bowel disease undergoing surveillance colonoscopy.

  * Patients with Crohn's (L2/L3 Montreal classification) with >50% colonic involvement
  * Patients with ulcerative colitis with Extensive or left sided disease (E3 or E2 Montreal classification) for at least 8 years or a diagnosis of Primary sclerosing cholangitis concomitant with IBD.

Exclusion Criteria:

* The participant may not enter the study if ANY of the following apply:

  * Disease duration <8 years unless a diagnosis of PSC
  * Incomplete colonoscopy
  * BBPS <6 or <2 in any segment
  * MES ≥2 or any variable of the SES-CD is ≥2 or any stenosis for >10cm segment (above the rectum)
  * Previous colorectal resection
  * Thrombocytopaenia (platelet count <50) or Coagulopathy precluding biopsy
  * Anticoagulation that has not been held appropriately prior to the procedure (must be held at least the morning of the procedure).
  * Allergy to Indigo Carmine
  * Pregnancy
  * Unable or unwilling to consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
To compare the proportion of patients with at least 1 dysplastic lesion detected using TXI compared with dye chromoendoscopy | 6 months
  The number of dysplastic areas detected during endoscopy

IPD SHARING:
Plan to Share IPD: No